CLINICAL TRIAL: NCT04956341
Title: Auricular Acupuncture for Sleep Disturbances: A Randomized Control Trial
Brief Title: Auricular Acupuncture for Sleep Disturbances
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FWH20210106H
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbance
Keywords: acupuncture; auricular acupuncture; sleep
MeSH Terms: conditions — Parasomnias | interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: At Visit 10 (final visit), those in the non-acupuncture group still experiencing symptoms will be offered the opportunity to be rolled into the acupuncture treatment arm of the study as outlined above. This will not be part of the analysis. If a patient in the acupuncture group is still having symptoms they will be referred back to their primary care manager for further evaluation at the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard treatment from PCM or Mental Health or both + auricular acupuncture (Experimental)
  Interventions: Device: Auricular acupuncture
- Standard treatment from Primary Care Manager (PCM) or Mental Health or both (Placebo Comparator)
  Interventions: Other: Standard treatment

INTERVENTIONS:
Device: Auricular acupuncture — Auricular acupuncture treatments will be utilizing ASP needles. The needles will stay in and fall out on their own (usually 3-10 days). For some patients who are acupuncture naïve, Seirin 15mm needles will be placed and allowed to remain for 45 minutes. This option will be provided to all subjects for their first treatment. Auricular acupuncture treatment possible locations will be as defined as: Master Cerebral/Prefrontal cortex, Amygdala, Hippocampus, Hypothalamus, Point Zero, Shen Men, Insomnia 1,Insomnia 2 OR Prefrontal Cortex, Reticular formation, Pineal gland, Hypothalamus, Point zero. In acupuncture parlance, the patient will be treated with ATP plus sleep I on first visit, then the acupuncturist will continue to use that treatment for each subsequent visit with the potential to add ATP plus sleep II. Both ears will be treated unless the patient requests that one be left open. The acupuncturist may use sleep I in one ear and sleep II in the other.
  Arms: Standard treatment from PCM or Mental Health or both + auricular acupuncture
Other: Standard treatment — Standard treatment from Primary Care Manager (PCM) or Mental Health or both
  Arms: Standard treatment from Primary Care Manager (PCM) or Mental Health or both

SUMMARY:
A randomized controlled trial of auricular acupuncture for sleep disturbances.

* Objective 1: Evaluate the effectiveness of a specific protocol of auricular acupuncture in the treatment of sleep disturbance among active duty and otherDoD beneficiaries.
* Objective 2: Test whether a brief course of auricular acupuncture treatments among active duty and other DoD beneficiaries with sleep disturbance willalso decrease severity of anxiety, depression, pain and improve sleep and social functioning in subgroup analysis of subjects with known or newlydiagnosed mental health disorders (e.g., anxiety disorders, depression).
* Null Hypothesis: Auricular Acupuncture has no effect on sleep disturbance.
* Alternative Hypothesis: Auricular Acupuncture reduces sleep disturbance.

DETAILED DESCRIPTION:
Active duty members and DoD beneficiaries aged 18-80 years old and meeting the inclusion/exclusion criteria will be offered an opportunity to participate.They will be recruited from the clinics at 99MDG (Nellis AFB), 96MDG (Eglin AFB), and 375 MDG (Scott AFB). All of the below items are research-relatedunless marked as 'standard of care'. All visits will last approximately 30 minutes in length.

Screening Visit:

* Obtain and document signed Informed Consent document and HIPAA Authorization.
* Review past medical history to verify the inclusion/exclusion criteria
* We will record health care resource utilization to include Number of hospital or clinic visits (previous encounters) for sleep problems in the past 12 months
* Medication use (Sleep medications, stimulant medications, energy drinks at least once/week), co-morbidities, phone number, e-mail address, dateof birth, gender, race, ethnicity, highest education level, total number of children in household), Service characteristics (officer, enlisted, retired)(service branch), History of deployment (never deployed, previously deployed, number of deployments), Usual Work pattern (Day, night),
* Record whether the subject has a history of Obstructive Sleep Apnea (OSA) and whether it is treated or untreated. If treated, do they use aContinuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP) machine? If patient uses CPAP/BiPAP, do they use it atleast 70% of the time as reported by patient or CPAP/BiPAP recent data pull in medical record. These questions are asked due to a possiblerelationship between OSA and sleep disturbance (3); those who have OSA and do not use a CPAP or use one infrequently need to be accounted forso as to not to confound data analysis.
* PROMIS-16 Sleep-Related Impairment Scale

Randomization:

Subjects who score a medium or severe on the PROMIS-16 (T-Score greater than or equal to 60). Sleep-Related Impairment Scale will berandomized into one of two groups and the intervention will be performed. The investigators acknowledge that any of these standard treatmentsmay be shorter or longer in duration than the duration of the study. There is no additional risk to subjects for continuing to track their sleeppatterns and mental health scores on various instruments shorter or longer than standard of care treatments. Furthermore, this study is meant tobe a pragmatic trial-there are many evidence based and not evidence based treatments for sleep disturbance that are considered standard ofcare. We seek to allow any of these treatments to proceed and evaluate the addition of auricular acupuncture as it can be applied in a clinic setting:

* Group 1: Standard treatment from Primary Care Manager (PCM) or Mental Health or both
* Group 2: Standard treatment from PCM or Mental Health or both + auricular Acupuncture

Visit 1 (0 weeks may be same day as screening visit):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles.
* All subjects will be given a Couples Satisfaction Index-4 (CSI-4) business card and asked to have their closest family member/friend aged 18 yearsor older complete the questionnaire on Survey Monkey at Visit 1, Visit 8, and Visit 10 (the dates will be on the back of the CSI-4 business card).They will be asked to have the same person complete all 3 questionnaires during the study.
* All subjects will take the following questionnaires via study electronic device or paper:
* PROMIS-16 Sleep-Related Impairment Scale (PROMIS-16)
* Measure Yourself Medical Outcome Profile (MYMOP) Initial

Visit 2 (1 week):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles.

Visit 3 (2 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles.

Visit 4 (3 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles -placed, and the location of the needles for each treatment.
* All subjects will take the following questionnaires via study electronic device or paper:

  * PROMIS-16
  * MYMOP Follow Up

Visit 5 (5 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles for each treatment.

Visit 6 (7 Weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles for each treatment.

Visit 7 (9 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles for each treatment.

Visit 8 (11 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles for each treatment.
* All subjects will take the following questionnaires via study electronic device or paper:

  * PROMIS-16
  * MYMOP Follow Up
* Subjects will be reminded to have their closest family member/friend aged 18 years or older complete the on-line CSI-4 questionnaire on SurveyMonkey on the dates noted on the back of the CSI-4 Business Card. They will be given another CSI-4 business card, if needed.

Visit 9 (15 weeks):

* Subjects will receive study procedures according to their randomization group.
* For subjects in group 2, the Research Coordinator will record the name of the investigator performing the auricular acupuncture, the number ofASP acupuncture needles placed, and the location of the needles for each treatment.
* All subjects will take the following questionnaires via study electronic device or paper:

  * PROMIS-16
  * MYMOP Follow Up

Visit 10 (23-24 Weeks):

* All subjects will take the following questionnaires via study electronic device or paper:

  * PROMIS-16
  * MYMOP Follow Up
* Subjects will be reminded to have their closest family member/friend aged 18 years or older complete the on-line CSI-4 questionnaire on SurveyMonkey on the dates noted on the back of the CSI-4 Business Card. They will be given another CSI-4 business card, if needed.

CROSSOVER:

At Visit 10 (final visit), those in the non-acupuncture group still experiencing symptoms will be offered the opportunity to be rolled into theacupuncture treatment arm of the study as outlined above. This will not be part of the analysis. If a patient in the acupuncture group is still havingsymptoms they will be referred back to their primary care manager for further evaluation at the conclusion of the study.

All study subjects will receive a $100 gift card at the completion of the 24 weeks. Active Duty and GS employees (who are also DoD beneficiaries) mayalso receive a $100 gift card only upon completion of the appropriate off-duty employment paperwork with their supervisor

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female Active Duty members and DoD beneficiaries ages 18-80 with complaints of sleep disturbances.
* PROMIS-16 Sleep-Related Impairment Scale with a score of medium or severe (T-Score greater than or equal to 60).

Exclusion Criteria:

* Patients with OSA who are prescribed CPAP/BiPAP and either do not use it or use it <70% of time per patient report.
* Investigators seek to exclude individuals with sleep-related medical or psychiatric conditions that are so severe as to render these patients inappropriate for treatment in primary care or simple mental health without psychiatry oversight or that acupuncture cannot be expected to have an effect on (e.g., thyroid disease). Specifically, exclusion criteria will include:

  * Psychosis
  * Thyroid disease undergoing active adjustment of medication.Depression, with suicidality. (clinician judgment)
  * Greater than 10 mg equivalent of diazepam equivalent per day for any reason
  * Non-response to greater than 2 PSTD treatments
* Having acupuncture not related to sleep in the past 3 months
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep-Related Impairment Scale | baseline, pre-intervention
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 1 (0 weeks/same day as screening)
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 2 (1 week) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 3 (2 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 4 (3 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 5 (5 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 6 (7 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 7 (9 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 8 (11 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 9 (15 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
PROMIS Sleep-Related Impairment Scale | visit 10 (23-24 weeks) post study visit procedures appropriate to subject randomization group
  Computer Adaptive Test (CAT) version OR The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. As additional items from the 16-item bank are administered, the potential for error is reduced and confidence in the respondent's score increases. CAT will continue until either the standard error drops below a specified level (on the T-score metric 3.0 for adult and adult cancer CATs), or the participant has answered the maximum number of questions (12), whichever occurs first.
  Sleep Related Impairment- Short form 8a (paper version). Subjects must answer all items (questions/statements) presented for a valid score
Measure Yourself Medical Outcome Profile (MYMOP) Initial | visit 1 (0 weeks)
  MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1.
Measure Yourself Medical Outcome Profile (MYMOP) Follow-up | visit 4 (3 weeks)
  MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1.
Measure Yourself Medical Outcome Profile (MYMOP) Follow-up | visit 8 (11 weeks)
  MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1.
Measure Yourself Medical Outcome Profile (MYMOP) Follow-up | visit 9 (15 weeks)
  MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1.
Measure Yourself Medical Outcome Profile (MYMOP) Follow-up | visit 10 (23-24 weeks)
  MYMOP employs a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score. Normative values are neither available nor meaningful for the MYMOP as it is individual to each patient; however, a clinically meaningful change is considered to be a change in the scores of more than 1.

SECONDARY OUTCOMES:
Couples Satisfaction Index CSI) | visit 1 (0 weeks)
  The CSI-4 is family member survey. CSI-4 scores can range from 0 to 21 and scores can be treated as a continuous variable. Higher scores indicate higher levels of relationship satisfaction. CSI-4 scores falling below 13.5 suggest notable relationship dissatisfaction.
  All subjects will be given a Couples Satisfaction Index-4 (CSI-4) business card and asked to have their closest family member/friend aged 18 years or older complete the questionnaire on Survey Monkey.
Couples Satisfaction Index CSI) | visit 8 (11 weeks)
  The CSI-4 is family member survey. CSI-4 scores can range from 0 to 21 and scores can be treated as a continuous variable. Higher scores indicate higher levels of relationship satisfaction. CSI-4 scores falling below 13.5 suggest notable relationship dissatisfaction.
  All subjects will be given a Couples Satisfaction Index-4 (CSI-4) business card and asked to have their closest family member/friend aged 18 years or older complete the questionnaire on Survey Monkey.
Couples Satisfaction Index CSI) | visit 10 (23-24 weeks)
  The CSI-4 is family member survey. CSI-4 scores can range from 0 to 21 and scores can be treated as a continuous variable. Higher scores indicate higher levels of relationship satisfaction. CSI-4 scores falling below 13.5 suggest notable relationship dissatisfaction.
  All subjects will be given a Couples Satisfaction Index-4 (CSI-4) business card and asked to have their closest family member/friend aged 18 years or older complete the questionnaire on Survey Monkey.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crawford, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Engel CC, Cordova EH, Benedek DM, Liu X, Gore KL, Goertz C, Freed MC, Crawford C, Jonas WB, Ursano RJ. Randomized effectiveness trial of a brief course of acupuncture for posttraumatic stress disorder. Med Care. 2014 Dec;52(12 Suppl 5):S57-64. doi: 10.1097/MLR.0000000000000237. PMID 25397825
- [Background] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Background] A Caldwell J, Knapik JJ, Lieberman HR. Trends and factors associated with insomnia and sleep apnea in all United States military service members from 2005 to 2014. J Sleep Res. 2017 Oct;26(5):665-670. doi: 10.1111/jsr.12543. Epub 2017 Apr 27. PMID 28448689
- [Background] Colvonen PJ, Straus LD, Stepnowsky C, McCarthy MJ, Goldstein LA, Norman SB. Recent Advancements in Treating Sleep Disorders in Co-Occurring PTSD. Curr Psychiatry Rep. 2018 Jun 21;20(7):48. doi: 10.1007/s11920-018-0916-9. PMID 29931537
- [Background] Troxel WM, Shih RA, Pedersen ER, Geyer L, Fisher MP, Griffin BA, Haas AC, Kurz J, Steinberg PS. Sleep in the Military: Promoting Healthy Sleep Among U.S. Servicemembers. Rand Health Q. 2015 Nov 30;5(2):19. eCollection 2015 Nov 30. PMID 28083395
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] National Institutes of Health. National Institutes of Health State of the Science Conference statement on Manifestations and Management of Chronic Insomnia in Adults, June 13-15, 2005. Sleep. 2005 Sep;28(9):1049-57. doi: 10.1093/sleep/28.9.1049. No abstract available. PMID 16268373
- [Background] Kulka RA, Schlenger WE, Fairbank JA, et al. Trauma and the Vietnam War Generation: Report of Findings From the National Vi etnam VeteransReadjustment Study. New York, NY: Brunner/Mazel; 1990.
- [Background] Margolies SO, Rybarczyk B, Vrana SR, Leszczyszyn DJ, Lynch J. Efficacy of a cognitive-behavioral treatment for insomnia and nightmares in Afghanistan and Iraq veterans with PTSD. J Clin Psychol. 2013 Oct;69(10):1026-42. doi: 10.1002/jclp.21970. Epub 2013 Apr 29. PMID 23629959
- [Background] Gellis, Les A., and Philip R. Gehrman, "Cognitive Behavioral Treatment for Insomnia in Veterans with Long-Standing Posttraumatic Stress Disorder: A Pilot Study," Journal of Aggression, Maltreatment and Trauma, Vol. 20, No. 8, 2011
- [Background] Brown CA, Berry R, Schmidt A. Sleep and military members: emerging issues and nonpharmacological intervention. Sleep Disord. 2013;2013:160374. doi: 10.1155/2013/160374. Epub 2013 Jul 14. PMID 23956864
- [Background] Talbot LS, Maguen S, Metzler TJ, Schmitz M, McCaslin SE, Richards A, Perlis ML, Posner DA, Weiss B, Ruoff L, Varbel J, Neylan TC. Cognitive behavioral therapy for insomnia in posttraumatic stress disorder: a randomized controlled trial. Sleep. 2014 Feb 1;37(2):327-41. doi: 10.5665/sleep.3408. PMID 24497661
- [Background] Koffel E, Farrell-Carnahan L. Feasibility and preliminary real-world promise of a manualized group-based cognitive behavioral therapy for insomnia protocol for veterans. Mil Med. 2014 May;179(5):521-8. doi: 10.7205/MILMED-D-13-00455. PMID 24806497
- [Background] Marmar CR, Schlenger W, Henn-Haase C, Qian M, Purchia E, Li M, Corry N, Williams CS, Ho CL, Horesh D, Karstoft KI, Shalev A, Kulka RA. Course of Posttraumatic Stress Disorder 40 Years After the Vietnam War: Findings From the National Vietnam Veterans Longitudinal Study. JAMA Psychiatry. 2015 Sep;72(9):875-81. doi: 10.1001/jamapsychiatry.2015.0803. PMID 26201054
- [Background] Neylan TC, Marmar CR, Metzler TJ, Weiss DS, Zatzick DF, Delucchi KL, Wu RM, Schoenfeld FB. Sleep disturbances in the Vietnam generation: findings from a nationally representative sample of male Vietnam veterans. Am J Psychiatry. 1998 Jul;155(7):929-33. doi: 10.1176/ajp.155.7.929. PMID 9659859
- [Background] Engdahl B, Dikel TN, Eberly R, Blank A Jr. Posttraumatic stress disorder in a community group of former prisoners of war: a normative response to severe trauma. Am J Psychiatry. 1997 Nov;154(11):1576-81. doi: 10.1176/ajp.154.11.1576. PMID 9356567
- [Background] Bei B, Asarnow LD, Krystal A, Edinger JD, Buysse DJ, Manber R. Treating insomnia in depression: Insomnia related factors predict long-term depression trajectories. J Consult Clin Psychol. 2018 Mar;86(3):282-293. doi: 10.1037/ccp0000282. PMID 29504795
- [Background] Mason EC, Harvey AG. Insomnia before and after treatment for anxiety and depression. J Affect Disord. 2014 Oct;168:415-21. doi: 10.1016/j.jad.2014.07.020. Epub 2014 Jul 18. PMID 25108278
- [Background] Mittal D, Drummond KL, Blevins D, Curran G, Corrigan P, Sullivan G. Stigma associated with PTSD: perceptions of treatment seeking combat veterans. Psychiatr Rehabil J. 2013 Jun;36(2):86-92. doi: 10.1037/h0094976. PMID 23750758
- [Background] Van Camp RO. Zolpidem in fatigue management for surge operations of remotely piloted aircraft. Aviat Space Environ Med. 2009 Jun;80(6):553-5. doi: 10.3357/asem.2460.2009. PMID 19522366
- [Background] King HC, Spence DL, Hickey AH, Sargent P, Elesh R, Connelly CD. Auricular acupuncture for sleep disturbance in veterans with post-traumatic stress disorder: a feasibility study. Mil Med. 2015 May;180(5):582-90. doi: 10.7205/MILMED-D-14-00451. PMID 25939115
- [Background] Grant S, Colaiaco B, Motala A, Shanman RM, Sorbero ME, Hempel S. Needle acupuncture for posttraumatic stress disorder (PTSD): A systematicreview. Santa Monica, CA: RAND Corporation, 15 March 2017.i-xxii, 1-94 pp. 2017:i-xxii, 1-94.
- [Background] King CH, Moore LC, Spence CD. Exploring Self-Reported Benefits of Auricular Acupuncture Among Veterans With Posttraumatic Stress Disorder. J Holist Nurs. 2016 Sep;34(3):291-9. doi: 10.1177/0898010115610050. Epub 2015 Nov 3. PMID 26530240
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Connor KM, Davidson JR. SPRINT: a brief global assessment of post-traumatic stress disorder. Int Clin Psychopharmacol. 2001 Sep;16(5):279-84. doi: 10.1097/00004850-200109000-00005. PMID 11552771
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Hou Y, Liu L, Chen X, Li Q, Li J. Association between circadian disruption and diseases: A narrative review. Life Sci. 2020 Dec 1;262:118512. doi: 10.1016/j.lfs.2020.118512. Epub 2020 Sep 30. PMID 33010281
- [Background] Leso V, Gervetti P, Mauro S, Macrini MC, Ercolano ML, Iavicoli I. Shift work and migraine: A systematic review. J Occup Health. 2020 Jan;62(1):e12116. doi: 10.1002/1348-9585.12116. PMID 32515906
- [Background] Oosterman JE, Wopereis S, Kalsbeek A. The Circadian Clock, Shift Work, and Tissue-Specific Insulin Resistance. Endocrinology. 2020 Dec 1;161(12):bqaa180. doi: 10.1210/endocr/bqaa180. PMID 33142318
- [Background] Smyth A, Jenkins M, Dunham M, Kutzer Y, Taheri S, Whitehead L. Systematic review of clinical practice guidelines to identify recommendations for sleep in type 2 diabetes mellitus management. Diabetes Res Clin Pract. 2020 Dec;170:108532. doi: 10.1016/j.diabres.2020.108532. Epub 2020 Nov 4. PMID 33157114
- [Background] Mohd Azmi NAS, Juliana N, Mohd Fahmi Teng NI, Azmani S, Das S, Effendy N. Consequences of Circadian Disruption in Shift Workers on Chrononutrition and their Psychosocial Well-Being. Int J Environ Res Public Health. 2020 Mar 19;17(6):2043. doi: 10.3390/ijerph17062043. PMID 32204445
- [Background] Kang J, Noh W, Lee Y. Sleep quality among shift-work nurses: A systematic review and meta-analysis. Appl Nurs Res. 2020 Apr;52:151227. doi: 10.1016/j.apnr.2019.151227. Epub 2019 Dec 26. PMID 31902652
- [Background] Jarnefelt H, Harma M, Sallinen M, Virkkala J, Paajanen T, Martimo KP, Hublin C. Cognitive behavioural therapy interventions for insomnia among shift workers: RCT in an occupational health setting. Int Arch Occup Environ Health. 2020 Jul;93(5):535-550. doi: 10.1007/s00420-019-01504-6. Epub 2019 Dec 18. PMID 31853633
- [Background] Moore BA, Tison LM, Palacios JG, Peterson AL, Mysliwiec V. Incidence of insomnia and obstructive sleep apnea in active duty United States military service members. Sleep. 2021 Jul 9;44(7):zsab024. doi: 10.1093/sleep/zsab024. PMID 33532830